CLINICAL TRIAL: NCT02537275
Title: Effect of the Pigment-free Optical Zone Diameter of Decorative Tinted Soft Contact Lenses on Visual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1-2014-0024
Record Dates: First submitted 2015-08-20; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Tinted Contact Lense

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- wearing contact lense group (Experimental): normal subjects after wearing tinted/normal contact lenses
  Interventions: Device: EyeLIKe Callamatch II, Koryo Eyetech Co, Seoul, Korea; Device: EyeLIKe Shine, Koryo Eyetech Co

INTERVENTIONS:
Device: EyeLIKe Callamatch II, Koryo Eyetech Co, Seoul, Korea — tinted contact lens, daily-wear tinted lens
Device: EyeLIKe Shine, Koryo Eyetech Co — clear lens

SUMMARY:
Investigators planned to investigate changes in visual function after wearing decorative tinted soft contact lenses with different pigment-free optical zone diameters.

ELIGIBILITY:
Inclusion Criteria:

* normal subject
* aged above 20 years old

Exclusion Criteria:

* subject who had a history of ocular diseases, such as ocular infection, ocular allergy, and autoimmune disease,
* patients with continuous use of topical ocular medications before surgery, or histories of ocular surgery or ocular injury.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
score of best-corrected visual acuity (BCVA) | 1 day

SECONDARY OUTCOMES:
Total score of ocular higher-order aberrations | 1 day
  ocular higher-order aberrations measured by iTrace (Tracey Technologies, Houston, Texas, USA; software V.4.1.0)
contrast sensitivity with tinted lense | 1 day
  contrast sensitivity measured by Optec 6500 test system (Stereo Optical Co, Chicago, Illinois, USA) at five spatial frequencies (1.5, 3, 6, 12 and 18 cycles/degree (cpd)) under photopic (luminance value of 85 candelas/square metre (cd/m2)) and mesopic conditions (target luminance value of 3 cd/m2) with or without glare after wearing clear lens and tinted lenses with different pigment-free optical zone diameters (4, 5 and 6 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Jung JW, Kim SM, Han SH, Kim EK, Seo KY, Kim TI. Effect of the pigment-free optical zone diameter of decorative tinted soft contact lenses on visual function. Br J Ophthalmol. 2016 May;100(5):633-7. doi: 10.1136/bjophthalmol-2015-306731. Epub 2015 Sep 16. PMID 26377415